CLINICAL TRIAL: NCT03450616
Title: Pilot Study Comparing Negative Pressure Dressings to Conventional Dressings for the Management of Patients With Venous Stasis Ulcers.
Brief Title: Pilot Study Comparing Negative Pressure Dressings to Conventional Dressings
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to begin study due to funding. PI has left organization
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-0951
Record Dates: First submitted 2018-02-23; First posted 2018-03-01 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Intervention Model Description: All subjects will receive both treatment arms at the same time.
Who Masked: Participant, Care Provider
Masking Description: Subjects and treating physician will be blinded to treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Negative Pressure Wound Therapy (Experimental): Subjects will have one venous stasis ulcer treated with the PICO Negative Pressure Wound Therapy Device
  Interventions: Device: PICO Negative Pressure Wound Therapy
- Compression Dressing- Standard of Care (Active Comparator): Subjects will have one venous stasis ulcer treated with the standard of care compression dressing.
  Interventions: Procedure: Compression Dressing

INTERVENTIONS:
Device: PICO Negative Pressure Wound Therapy — Negative Pressure Wound Therapy Device
  Arms: Negative Pressure Wound Therapy
Procedure: Compression Dressing — Standard of Care Compression Dressing
  Arms: Compression Dressing- Standard of Care

SUMMARY:
This study is being conducted to determine how the PICO™ Negative Pressure Wound Therapy compares to standard care treatment for venous stasis ulcers, as there is no evidence to date.

DETAILED DESCRIPTION:
This is a single-blind, randomized pilot study conducted in patients with bilateral venous stasis leg ulcers.

The aim of the study is to compare the rate of healing for venous stasis ulcers when using the PICO™ single use Negative pressure wound therapy (NPWT) system versus standard care.

The primary objective is to determine if the PICO™ NPWT system results in an increased rate of healing when compared to standard of care for the treatment of venous stasis ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Patient with bilateral venous leg ulcers (one on each lower extremity) (defined as any break in the skin that has either been present for longer than 6 wks or occurred in a person with a history of venous leg ulceration).
* The ulcer is required to be venous in appearance (ie: moist, shallow, and of an irregular shape), and judged unlikely to heal within 21 days.
* 18 years old or older
* Have an ankle brachial pressure index of at least 0.8 that was measured within the previous 3 months.

Exclusion Criteria:

* • Patients on anticoagulants- (ie: warfarin, direct thrombin inhibitors).

  * Patients who have a pressure index measured within the previous 3 months to be greater than 1.20
  * Patients with venous stasis ulcers greater than 17cm by 17cm.
  * Gross leg edema
  * Severe wound exudate
  * Patients with malignancy in the wound bed or margins of the wound
  * Previously confirmed and untreated osteomyelitis.
  * Patients with necrotic tissue with eschar present.
  * Patients with wounds that involve exposed arteries, veins, nerves, bone fragments or sharp edges.
  * Patients with wounds that requires surgical suction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Rate of healing | Weekly for three weeks
  Surface area and depth of wound measurements will be collected to determine rate of healing

CONTACTS AND LOCATIONS:
Locations (1):
- Staten Island University Hospital, Staten Island, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be made available to other researchers.